CLINICAL TRIAL: NCT02024425
Title: A Randomized, Double-blind Trial to Evaluate the Effect of a Functional Bioactive Supplement Associated With a Hypocaloric Equilibrated Diet to Treatment of Obese and Overweight Individuals
Brief Title: Functional Bioactive Supplement Effect in Lost Weight Treatment
Acronym: ALIBIRDII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALIBIRDII
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Obesity and Overweight
Keywords: Clinical trials; Adult; Women; Functional food; Dietary Supplements; Overweight; Obese; Absorptiometry, Dual X-Ray; Rosmarinus; Oligosaccharides; Lactulose; Bioactive peptide
MeSH Terms: conditions — Obesity; Overweight | interventions — Antioxidants; Oligosaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional bioactive supplement (Active Comparator): The functional bioactive supplement is composed of antioxidant extracted from rosemary, oligosaccharides derived from lactulose and bioactive peptides. It will be used for obese and overweight treatment
  Interventions: Dietary Supplement: Functional bioactive supplement
- Maltodextrin and saccharose (Placebo Comparator): The control supplement is composed of maltodextrin and saccharose . It has no effect for obese and overweight treatment
  Interventions: Dietary Supplement: Control supplement

INTERVENTIONS:
Dietary Supplement: Functional bioactive supplement — 1,25g of antioxidant extracted from rosemary, 18g of oligosaccharides derived from lactulosa and 1,25g of bioactive peptides
  Other Names: antioxidant, oligosaccharides and bioactive peptides
  Arms: Functional bioactive supplement
Dietary Supplement: Control supplement
  Arms: Maltodextrin and saccharose

SUMMARY:
The purpose this study is to evaluate the therapeutic effect of a functional bioactive supplement associated with a hypocaloric equilibrated diet to treat obese and overweight individuals. The functional bioactive supplement, containing antioxidant extracted from rosemary, oligosaccharides derived from lactulose and bioactive peptides, was developed to satiety control, improves of anti-inflammatory response and antioxidant defense mechanisms as well as to weight loss.

DETAILED DESCRIPTION:
A randomized, parallel, double-blind, controlled was performed to evaluate the therapeutic effect of a functional bioactive supplement associated with a hypocaloric equilibrated diet to treatment of obesity and overweight.

Women aged between 18 and 65 years with obesity and overweight diagnosis (IMC >25<35 kg/m2) were included in the study. The clinical trial will be performed in the Clinical Nutrition Department of La Paz University Hospital, in Madrid. All of the volunteers will receive a dietetic treatment with 1500 Kcal/day and physical activity recommendations during the study.

ELIGIBILITY:
Inclusion Criteria:

* Women from 45 to 75 years old;
* Overweight (IMC ≥25<30 Kg/m2) or obese (IMC ≥30<35 Kg/m2) volunteers
* Signed informed consent.

Exclusion Criteria:

* Subjects with drug consumption (lipid-lowering, oral hypoglycemic agents and / or hypertensive) in less than one month period;
* Subjects with Diabetes Mellitus insulin dependent;
* Individuals that stop smoking in the next 12 weeks (during the study);
* Subjects with increased alcohol consumption (> 1 glass of vine);
* Subjects that consume drugs, vitamins, minerals, prebiotics or/and probiotics that interfere with the body's response to the extracts in the 2 weeks before to baseline;
* Subjects with drugs consumption special diet due to disease as celiac disease, chronic renal failure, etc;
* Subjects with disorders associated with eating behaviour;
* Subjects with drugs or supplements consumption to weight lost;
* Subjects with physical problems complying with the recommendations of physical activity and diet indicated;
* Subjects who refuse to perform the indicated dietary changes throughout the study;
* Subjects with diseases that could be involucrate in weight lost (not controlled hypothyroidism, serious psychiatric illness, etc.);
* Subjects with mental disease or low cognitive function;
* Subjects with severe diseases (hepatic, kidney, cancer…);
* Pregnant women or lactating;
* Subjects with physical problems complying with the recommendations of physical activity.
* Subjects with intensive physical activity;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | 12 weeks
  Clinical response - changes in body composition: weight, waist circumference and Absorptiometry, Dual X-Ray.The primary outcome result measurement was the lost weight, changes in body composition

SECONDARY OUTCOMES:
Life style and health status: Life style and physical activity questionnaire | Week 0 and Week 12
Genetic analysis | Week 0 and Week 12
Metabolomic analyses | Week 0 and Week 12
Endothelial function markers | Week 0 y Week 12
  Endothelial function markers: eNOS, VCAM-1, PAI1 and blood pressure
Satiety hormones | Week 0 y Week 12
  Satiety hormones: ghrelin, GLP-1; Leptin; adiponectin and NPY
Inflammatory markers | Week 0 and Week 12
  Inflammatory markers: TNF-α, IL-6, PCR and fibrinogen
Glucose Metabolism | Week 0 and Week 12
  Glucose Metabolism: glucose, basal insulin, HbA1c (in diabetic patients), HOMA index (glycemic insulin sensitivity index was calculated using the formula: HOMA-IR = fasting glucose (mmol/l)/fasting immunoreactive insulin (mU/ml)/22•5)
Lipid profile: Cholesterol | Week 0 and Week 12
  Lipid profile: Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides
Oxidative Stress Parameters | Week 0 and Week 12
  Oxidative Stress Parameters: plasma antioxidant capacity (FRAP, ferric reducing antioxidant power) and lipidic peroxidation (TBARS, thiobarbituric acid reactive substances assay), oxidized LDL, PON1, F2-isoprostanes
Adverse effects | 0 , 3, 6, 9 and 12 weeks
  Adverse effects: transaminases and creatinine

OTHER OUTCOMES:
Appetite and satiety | 0 , 3, 6, 9 and 12 weeks
Frequent daily evacuations | 4 Weeks
  Frequent daily evacuations, format and consistency of the feces, total and segmental transit time. The format and consistency of the feces was evaluated in accordance with the Bristol Stool Form Scale (stool are rated based on water content of the feces, with 1 meaning hard stools to 7 meaning liquid stools)
Adherence and Tolerance Parameters | 0 , 3, 6, 9 and 12 weeks
  Adherence and Tolerance Parameters: adherence and tolerance to the products and diet prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gomez Candela, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- See also: Institute for Health Research IdiPAZ — http://www.idipaz.es